CLINICAL TRIAL: NCT02850653
Title: Contribution of Fast Molecular Bacterial Identification by Real-time PCR in Managing of Postoperative Acute Endophthalmitis
Brief Title: Targeted PCR and Acute Endophthalmitis
Acronym: Targeted PCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC07.006
Record Dates: First submitted 2016-07-11; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Acute Endophthalmitis Post-operative
Keywords: Acute Endophthalmitis.; PCR; Ocular sampling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endophthalmitis sufferers (Other): Patients hospitalized for diagnostic and therapeutic evaluation of a post-operative acute endophthalmitis.
  Interventions: Biological: PCR : 16S ribosomal DNA and real-time targeted PCR; Biological: Sampling of aqueous humour
- Healthy control patient (Other): Patients hospitalized in the context of a scheduled surgery with sampling of aqueous humour.
  Interventions: Biological: PCR : 16S ribosomal DNA and real-time targeted PCR; Biological: Sampling of aqueous humour

INTERVENTIONS:
Biological: PCR : 16S ribosomal DNA and real-time targeted PCR
Biological: Sampling of aqueous humour

SUMMARY:
Endophthalmitis is a serious eye infection of exogenous origin (post-operational, post-traumatic) or endogenous origin (metastatic). This is a diagnostic and therapeutic emergency.

Each patient suffering from endophthalmitis must have immediately an ocular sampling, an intra ocular injection of antibiotics and a systemic antibiotic cover.

The etiological treatment will be adapted according to the infectious agent.

DETAILED DESCRIPTION:
The main goal of this prospective multi-centre trial is to improve the sensitivity and rapidity of the infectious agent's identification involved in endophthalmitis cases, particularly virulent species (like Staphylococcus aureus, Streptococcus pneumoniae...) from ocular samples with the help of real-time PCR.

This will help the ophthalmologist to be more efficient in accordance with the kind of the bacteria.

Data will also enable to compare both PCR techniques used in this study. The secondary goal of the prospective study is to characterize the resistance of bacterial's species found during acute endophthalmitis with the antibiogram and by the study of resistance genes, to enable to correlate the resistance in vitro with the therapeutic response in vivo and get precious epidemiological data to adapt prophylactic antibiotic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects affiliated to the social security system
* Signed informed consent documentation
* Patients over 18 years
* Male or female person
* Patients hospitalized for diagnostic and therapeutic evaluation of a post-operative acute endophthalmitis, or within the context of a scheduled surgery with sampling of aqueous humour.
* Has given his or her consent, having been provided with detailed informations regarding to intraocular sampling.

Exclusion Criteria:

* antibiotherapy via intravenous (< 8 days) for patients NON suffering from endophthalmitis (control group)
* Patient's participation to the study refused
* Patients under 18 years
* Patients adults under guardianship or curatorship, or unable to express his/her consent.
* Pregnant women
* Breastfeeding women
* Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Visual acuteness | 2 minutes
  Clinical follow-up of patients
Intraocular pressure | 5 minutes
  Clinical follow-up of patients
Biomicroscopic exam with the slit lamp | 3 minutes
  State of anterior and posterior segment (back of the eye)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Chiquet, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Microbiologic factors and visual outcome in the endophthalmitis vitrectomy study. Am J Ophthalmol. 1996 Dec;122(6):830-46. doi: 10.1016/s0002-9394(14)70380-0. PMID 8956638
- [Background] Adam D. Global antibiotic resistance in Streptococcus pneumoniae. J Antimicrob Chemother. 2002 Jul;50 Suppl:1-5. doi: 10.1093/jac/dkf801. PMID 12077153
- [Background] Alexandrakis G, Alfonso EC, Miller D. Shifting trends in bacterial keratitis in south Florida and emerging resistance to fluoroquinolones. Ophthalmology. 2000 Aug;107(8):1497-502. doi: 10.1016/s0161-6420(00)00179-2. PMID 10919897
- [Background] Anand AR, Madhavan HN, Therese KL. Use of polymerase chain reaction (PCR) and DNA probe hybridization to determine the Gram reaction of the infecting bacterium in the intraocular fluids of patients with endophthalmitis. J Infect. 2000 Nov;41(3):221-6. doi: 10.1053/jinf.2000.0731. PMID 11120608
- [Background] Ariyasu RG, Nakamura T, Trousdale MD, Smith RE. Intraoperative bacterial contamination of the aqueous humor. Ophthalmic Surg. 1993 Jun;24(6):367-73; discussion 373-4. PMID 8336886
- [Background] Auclin F, Pollet E, Roman S, Boureau-Andrieux C, Leroux-Les-Jardins S, Ullern M. [Fifty-two cases of postoperative endophthalmitis treated with one protocol: anatomical and functional results]. J Fr Ophtalmol. 2001 Sep;24(7):687-91. French. PMID 11591907
- [Background] Barry P, Seal DV, Gettinby G, Lees F, Peterson M, Revie CW; ESCRS Endophthalmitis Study Group. ESCRS study of prophylaxis of postoperative endophthalmitis after cataract surgery: Preliminary report of principal results from a European multicenter study. J Cataract Refract Surg. 2006 Mar;32(3):407-10. doi: 10.1016/j.jcrs.2006.02.021. PMID 16631047
- [Background] Benz MS, Scott IU, Flynn HW Jr, Unonius N, Miller D. Endophthalmitis isolates and antibiotic sensitivities: a 6-year review of culture-proven cases. Am J Ophthalmol. 2004 Jan;137(1):38-42. doi: 10.1016/s0002-9394(03)00896-1. PMID 14700642
- [Background] Blondeau JM. Fluoroquinolones: mechanism of action, classification, and development of resistance. Surv Ophthalmol. 2004 Mar;49 Suppl 2:S73-8. doi: 10.1016/j.survophthal.2004.01.005. PMID 15028482
- [Background] Bron A. [Endophthalmitis. 1: diagnosis]. J Fr Ophtalmol. 1996;19(3):225-40. No abstract available. French. PMID 8731774
- [Background] Carroll NM, Jaeger EE, Choudhury S, Dunlop AA, Matheson MM, Adamson P, Okhravi N, Lightman S. Detection of and discrimination between gram-positive and gram-negative bacteria in intraocular samples by using nested PCR. J Clin Microbiol. 2000 May;38(5):1753-7. doi: 10.1128/JCM.38.5.1753-1757.2000. PMID 10790093
- [Background] Chen CC, Teng LJ, Chang TC. Identification of clinically relevant viridans group streptococci by sequence analysis of the 16S-23S ribosomal DNA spacer region. J Clin Microbiol. 2004 Jun;42(6):2651-7. doi: 10.1128/JCM.42.6.2651-2657.2004. PMID 15184447
- [Background] Chiquet C, Creuzot-Garcher C, Rouberol F, Palombi K, Bron A, Denis P, Lafontaine PO, Benito Y, Cornut PL, Thuret G, Romanet JP, Vandenesch F. Bacterial identification using PCR in a large series of acute post-cataract endophthalmitis; 2006a; Vilamoura, Portugal
- [Background] Chiquet C, Lafontaine PO, Benito Y, Cornut PL, Palombi K, Thuret G, Creuzot-Garcher C, Denis P, Romanet JP, Vandenesch F. Bacterial identification using PCR in a large series of acute post-cataract endophthalmitis; 2006b; Fort Lauderdale, USA.
- [Background] Chiquet C, Lina G, Benito Y, Cornut PL, Etienne J, Romanet JP, Denis P, Vandenesch F. Polymerase chain reaction identification in aqueous humor of patients with postoperative endophthalmitis. J Cataract Refract Surg. 2007 Apr;33(4):635-41. doi: 10.1016/j.jcrs.2006.12.017. PMID 17397736
- [Background] Corless CE, Guiver M, Borrow R, Edwards-Jones V, Fox AJ, Kaczmarski EB. Simultaneous detection of Neisseria meningitidis, Haemophilus influenzae, and Streptococcus pneumoniae in suspected cases of meningitis and septicemia using real-time PCR. J Clin Microbiol. 2001 Apr;39(4):1553-8. doi: 10.1128/JCM.39.4.1553-1558.2001. PMID 11283086
- [Background] Cornut PL, Chiquet C, Bron A, Romanet JP, Lina G, Lafontaine PO, Benito Y, Pechinot A, Burillon C, Vandenesch F, Denis P; FRIENDS Group. Microbiologic identification of bleb-related delayed-onset endophthalmitis caused by moraxella species. J Glaucoma. 2008 Oct-Nov;17(7):541-5. doi: 10.1097/IJG.0b013e31816299ec. PMID 18854730
- [Background] D'Amico DJ. 2000. Principles and Practice of Ophthalmology - Postoperative endophthalmitis
- [Background] Dickey JB, Thompson KD, Jay WM. Anterior chamber aspirate cultures after uncomplicated cataract surgery. Am J Ophthalmol. 1991 Sep 15;112(3):278-82. doi: 10.1016/s0002-9394(14)76728-5. PMID 1882939
- [Background] Egger SF, Huber-Spitzy V, Scholda C, Schneider B, Grabner G. Bacterial contamination during extracapsular cataract extraction. Prospective study on 200 consecutive patients. Ophthalmologica. 1994;208(2):77-81. doi: 10.1159/000310457. PMID 8183529
- [Background] Ferro JF, de-Pablos M, Logrono MJ, Guisasola L, Aizpuru F. Postoperative contamination after using vancomycin and gentamicin during phacoemulsification. Arch Ophthalmol. 1997 Feb;115(2):165-70. doi: 10.1001/archopht.1997.01100150167003. PMID 9046249
- [Background] Feys J, Emond JP, Salvanet-Bouccara A, Dublanchet A. [Bacteriological study of the intraocular fluid at the end of cataract surgery]. J Fr Ophtalmol. 1993;16(10):501-5. French. PMID 8301003
- [Background] Fisch A, Salvanet A, Prazuck T, Forestier F, Gerbaud L, Coscas G, Lafaix C. Epidemiology of infective endophthalmitis in France. The French Collaborative Study Group on Endophthalmitis. Lancet. 1991 Nov 30;338(8779):1373-6. PMID 1682746
- [Background] Gimbel HV, Sun R, DeBroff BM, Yang HM. Anterior chamber fluid cultures following phacoemulsification and posterior chamber lens implantation. Ophthalmic Surg Lasers. 1996 Feb;27(2):121-6. PMID 8640434
- [Background] Goldstein MH, Kowalski RP, Gordon YJ. Emerging fluoroquinolone resistance in bacterial keratitis: a 5-year review. Ophthalmology. 1999 Jul;106(7):1313-8. PMID 10406613
- [Background] Han DP, Wisniewski SR, Kelsey SF, Doft BH, Barza M, Pavan PR. Microbiologic yields and complication rates of vitreous needle aspiration versus mechanized vitreous biopsy in the Endophthalmitis Vitrectomy Study. Retina. 1999;19(2):98-102. doi: 10.1097/00006982-199902000-00002. PMID 10213233
- [Background] Han DP, Wisniewski SR, Wilson LA, Barza M, Vine AK, Doft BH, Kelsey SF. Spectrum and susceptibilities of microbiologic isolates in the Endophthalmitis Vitrectomy Study. Am J Ophthalmol. 1996 Jul;122(1):1-17. doi: 10.1016/s0002-9394(14)71959-2. PMID 8659579
- [Background] Hooper DC. Mechanisms of fluoroquinolone resistance. Drug Resist Updat. 1999 Feb;2(1):38-55. doi: 10.1054/drup.1998.0068. PMID 11504468
- [Background] Hwang DG. Fluoroquinolone resistance in ophthalmology and the potential role for newer ophthalmic fluoroquinolones. Surv Ophthalmol. 2004 Mar;49 Suppl 2:S79-83. doi: 10.1016/j.survophthal.2004.01.004. PMID 15028483
- [Background] Hykin PG, Tobal K, McIntyre G, Matheson MM, Towler HM, Lightman SL. The diagnosis of delayed post-operative endophthalmitis by polymerase chain reaction of bacterial DNA in vitreous samples. J Med Microbiol. 1994 Jun;40(6):408-15. doi: 10.1099/00222615-40-6-408. PMID 8006933
- [Background] Jaeger EE, Carroll NM, Choudhury S, Dunlop AA, Towler HM, Matheson MM, Adamson P, Okhravi N, Lightman S. Rapid detection and identification of Candida, Aspergillus, and Fusarium species in ocular samples using nested PCR. J Clin Microbiol. 2000 Aug;38(8):2902-8. doi: 10.1128/JCM.38.8.2902-2908.2000. PMID 10921948
- [Background] Knox CM, Cevallos V, Margolis TP, Dean D. Identification of bacterial pathogens in patients with endophthalmitis by 16S ribosomal DNA typing. Am J Ophthalmol. 1999 Oct;128(4):511-2. doi: 10.1016/s0002-9394(99)00181-6. PMID 10577597
- [Background] Koc F, Akcam Z, Kuruoglu S, Oge I, Gunaydin M. Does surgical technique influence cataract surgery contamination? Eur J Ophthalmol. 2001 Jan-Mar;11(1):31-6. doi: 10.1177/112067210101100107. PMID 11284482
- [Background] Kohn AN. Bacterial cultures of lenses removed during cataract surgery. Am J Ophthalmol. 1978 Aug;86(2):162-6. doi: 10.1016/s0002-9394(14)76805-9. PMID 308320
- [Background] Koul S, Philipson A, Philipson BT. Incidence of endophthalmitis in Sweden. Acta Ophthalmol (Copenh). 1989 Oct;67(5):499-503. doi: 10.1111/j.1755-3768.1989.tb04099.x. PMID 2589048
- [Background] Lohmann CP, Heeb M, Linde HJ, Gabel VP, Reischl U. Diagnosis of infectious endophthalmitis after cataract surgery by polymerase chain reaction. J Cataract Refract Surg. 1998 Jun;24(6):821-6. doi: 10.1016/s0886-3350(98)80138-7. PMID 9642595
- [Background] Lohmann CP, Linde HJ, Reischl U. Improved detection of microorganisms by polymerase chain reaction in delayed endophthalmitis after cataract surgery. Ophthalmology. 2000 Jun;107(6):1047-51; discussion 1051-2. doi: 10.1016/s0161-6420(00)00083-x. PMID 10857821
- [Background] Mandelbaum S, Forster RK. 1996. Exogenous endophthalmitis. In: Pepose JS HGN, Wilhelmus K.R., editor. Ocular infection and Immunity: Mosby. p 1298-1320.
- [Background] Mistlberger A, Ruckhofer J, Raithel E, Muller M, Alzner E, Egger SF, Grabner G. Anterior chamber contamination during cataract surgery with intraocular lens implantation. J Cataract Refract Surg. 1997 Sep;23(7):1064-9. doi: 10.1016/s0886-3350(97)80081-8. PMID 9379378
- [Background] Oguz H, Satici A, Guzey M, Aslan G, Tasci S. Microbiologic analysis of aqueous humor in phacoemulsification. Jpn J Ophthalmol. 1999 May-Jun;43(3):162-5. doi: 10.1016/s0021-5155(99)00013-1. PMID 10413248
- [Background] Okhravi N, Adamson P, Carroll N, Dunlop A, Matheson MM, Towler HM, Lightman S. PCR-based evidence of bacterial involvement in eyes with suspected intraocular infection. Invest Ophthalmol Vis Sci. 2000 Oct;41(11):3474-9. PMID 11006241
- [Background] Okhravi N, Adamson P, Matheson MM, Towler HM, Lightman S. PCR-RFLP-mediated detection and speciation of bacterial species causing endophthalmitis. Invest Ophthalmol Vis Sci. 2000 May;41(6):1438-47. PMID 10798660
- [Background] Passemard M, Lafontaine PO, Pechinot A, Cornut PL, Rouberol F, Romanet JP, Bron A, Creuzot-Garcher C, Chiquet C. Antibiotic resistances of bacteria identified in an Endophthalmitis Prospective Study.; 2006; Fort lauderdale, USA.
- [Background] Pospisil A, Pospisil F, Dupont MJ, Delbosc B, Montard M. [Bacterial contamination of the anterior chamber and cataract surgery]. J Fr Ophtalmol. 1993;16(1):10-3. French. PMID 8482794
- [Background] Recchia FM, Busbee BG, Pearlman RB, Carvalho-Recchia CA, Ho AC. Changing trends in the microbiologic aspects of postcataract endophthalmitis. Arch Ophthalmol. 2005 Mar;123(3):341-6. doi: 10.1001/archopht.123.3.341. PMID 15767476
- [Background] Records RE, Iwen PC. Experimental bacterial endophthalmitis following extracapsular lens extraction. Exp Eye Res. 1989 Nov;49(5):729-37. doi: 10.1016/s0014-4835(89)80034-x. PMID 2591490
- [Background] Relman DA. 1993. Universal bacterial 16S rDNA amplification and sequencing. In: Persing DHea, editor. Diagnostic molecular microbiology Principles and applications. Washington, DC: ASM. p 489-495.
- [Background] Sakai H, Procop GW, Kobayashi N, Togawa D, Wilson DA, Borden L, Krebs V, Bauer TW. Simultaneous detection of Staphylococcus aureus and coagulase-negative staphylococci in positive blood cultures by real-time PCR with two fluorescence resonance energy transfer probe sets. J Clin Microbiol. 2004 Dec;42(12):5739-44. doi: 10.1128/JCM.42.12.5739-5744.2004. PMID 15583307
- [Background] Salvanet-Bouccara A, Forestier F, Coscas G, Adenis JP, Denis F. [Bacterial endophthalmitis. Ophthalmological results of a national multicenter prospective survey]. J Fr Ophtalmol. 1992;15(12):669-78. French. PMID 1299678
- [Background] Samson CM, Foster CS. 2002. Masquerades syndromes: endophthalmitis. In: A.T. FCSaV, editor. Diagnosis and treatment of uveitis. Philadelphia: WB Saunders. p 528-536.
- [Background] Seal DV, Barry P, Gettinby G, Lees F, Peterson M, Revie CW, Wilhelmus KR; ESCRS Endophthalmitis Study Group. ESCRS study of prophylaxis of postoperative endophthalmitis after cataract surgery: Case for a European multicenter study. J Cataract Refract Surg. 2006 Mar;32(3):396-406. doi: 10.1016/j.jcrs.2006.02.014. PMID 16631046
- [Background] Sobaci G, Tuncer K, Tas A, Ozyurt M, Bayer A, Kutlu U. The effect of intraoperative antibiotics in irrigating solutions on aqueous humor contamination and endophthalmitis after phacoemulsification surgery. Eur J Ophthalmol. 2003 Nov-Dec;13(9-10):773-8. doi: 10.1177/1120672103013009-1007. PMID 14700098
- [Background] Speaker MG, Milch FA, Shah MK, Eisner W, Kreiswirth BN. Role of external bacterial flora in the pathogenesis of acute postoperative endophthalmitis. Ophthalmology. 1991 May;98(5):639-49; discussion 650. doi: 10.1016/s0161-6420(91)32239-5. PMID 2062496
- [Background] Srinivasan R, Tiroumal S, Kanungo R, Natarajan MK. Microbial contamination of the anterior chamber during phacoemulsification. J Cataract Refract Surg. 2002 Dec;28(12):2173-6. doi: 10.1016/s0886-3350(02)01493-1. PMID 12498855
- [Background] Stefani S, Varaldo PE. Epidemiology of methicillin-resistant staphylococci in Europe. Clin Microbiol Infect. 2003 Dec;9(12):1179-86. doi: 10.1111/j.1469-0691.2003.00698.x. PMID 14686982
- [Background] Tervo T, Ljungberg P, Kautiainen T, Puska P, Lehto I, Raivio I, Jarvinen E, Kuusela P, Tarkkanen A. Prospective evaluation of external ocular microbial growth and aqueous humor contamination during cataract surgery. J Cataract Refract Surg. 1999 Jan;25(1):65-71. doi: 10.1016/s0886-3350(99)80013-3. PMID 9888079
- [Background] Therese KL, Anand AR, Madhavan HN. Polymerase chain reaction in the diagnosis of bacterial endophthalmitis. Br J Ophthalmol. 1998 Sep;82(9):1078-82. doi: 10.1136/bjo.82.9.1078. PMID 9893601
- [Background] Watanabe K, Numata-Watanabe K, Hayasaka S. Methicillin-resistant staphylococci and ofloxacin-resistant bacteria from clinically healthy conjunctivas. Ophthalmic Res. 2001 May-Jun;33(3):136-9. doi: 10.1159/000055659. PMID 11340403